CLINICAL TRIAL: NCT05389137
Title: To Identify the Immunogenicity and Safety of Inavtivated Quadrivalent Influenza Virus Split Vaccine in Children Aged 3-8 Years With Two Doses and One Dose Pre-immunization
Brief Title: To Identify the Immunogenicity and Safety of QIV in Children Aged 3-8 Years
Acronym: QIV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wuhan Institute of Biological Products Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: WIBP2021007
Record Dates: First submitted 2022-04-14; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: This clinical trial was designed as a self-controlled trial to observe the immunogenicity and safety. This study was an exploratory study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Trial group 1 (No previous influenza vaccination) (Other): Subjects with no previous influenza vaccination
  Interventions: Biological: Inavtivated Quadrivalent Influenza Virus Split Vaccine
- Trial group 2 (previous vaccinated with one dose of influenza vaccine) (Other): Subjects previously vaccinated with one dose of influenza vaccine
  Interventions: Biological: Inavtivated Quadrivalent Influenza Virus Split Vaccine
- Trial group 2 (previous vaccinated with two doses of influenza vaccine) (Other): Subjects previously vaccinated with two dose of influenza vaccine
  Interventions: Biological: Inavtivated Quadrivalent Influenza Virus Split Vaccine

INTERVENTIONS:
Biological: Inavtivated Quadrivalent Influenza Virus Split Vaccine — Prevent influenza caused by H1N1, H3N2, B (V), B (Y) strain virus infection.

SUMMARY:
To explore the immunogenicity and safety of quadrivalent split influenza virus vaccine in children aged 3-8 years with two doses and one dose. This clinical trial was designed as a self-controlled trial to observe the immunogenicity and safety. This study was an exploratory study.

Sample size and test grouping:

In this study, a total of 360 subjects were enrolled in a self-controlled trial design.

In this study, 360 subjects aged 3 to 8 years old were enrolled. According to their previous influenza vaccine vaccination status, they were assigned to experimental group 1 (no previous influenza vaccine), experimental group 2 (one dose of influenza vaccine previously) and experimental group 3 (two or more doses of influenza vaccine previously), with 120 cases in each experimental group.

All subjects received one dose of tetravalent influenza virus lysis vaccine on day 0,28 for immunogenicity and safety observation.

DETAILED DESCRIPTION:
Sample size and test grouping:

In this study, a total of 360 subjects were enrolled in a self-controlled trial design.

In this study, 360 subjects aged 3 to 8 years old were enrolled. According to their previous influenza vaccine vaccination status, they were assigned to experimental group 1 (no previous influenza vaccine), experimental group 2 (one dose of influenza vaccine previously) and experimental group 3 (two or more doses of influenza vaccine previously), with 120 cases in each experimental group.

All subjects received one dose of tetravalent influenza virus lysis vaccine on day 0,28 for immunogenicity and safety observation.

The enrollment sequence of this study is divided into two stages:

First stage: group 1, group 2 and group 3 into the group of 20 people, each agent 1 test vaccine respectively, collecting agent 1 test vaccine adverse event, within 7 days after 8 days after 1 dose diary collection card security assessment, confirm safe (not to suspend/terminate the test standard), can be on to the next stage into the group; The second dose of the trial vaccine was administered, adverse events were collected within 7 days after the second dose of the trial vaccine, diary cards were collected for safety assessment 8 days after the second dose, and the next phase of the second dose of vaccine could be administered after the safety was confirmed (criteria for suspension/termination of the trial were not met);

The second stage: The remaining 100 subjects in experimental groups 1, 2 and 3 were inoculated with the first and second doses of experimental vaccine.

Blood collection procedure:

About 4.0ml of venous blood was collected from all subjects before each dose and 30 days after the second dose.

ELIGIBILITY:
Inclusion Criteria:

1. At the age of 3 years old and below 9 years old on the day of enrollment, valid identification of the subject and/or his/her guardian can be provided;
2. The subject's guardian has the ability to understand the study requirements and process, agree to participate in the clinical trial and sign the informed consent (8-year-old subject: The subject and his/her guardian voluntarily agree to participate in the study, and the informed consent shall be signed by his/her guardian and the subject shall sign the informed consent for minors; Subjects aged 3-7: The guardian of the subject voluntarily agrees that the child should participate in the study, and the guardian should sign the informed consent);
3. The subject's guardian is competent to understand the study procedures, and the subject and/or his/her guardian are able to attend all planned follow-up visits;
4. Axillary temperature on the day of enrollment < 37.5℃.

Exclusion Criteria:

1. Have a history of severe allergy to any components of the test vaccine (including eggs and ovalbumin, etc.), such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, and local allergic necrosis reaction (Arthus reaction);
2. patients with influenza or influenza-like symptoms within 3 months (fever < axillary temperature ≥38℃ >, accompanied by cough or sore throat);
3. Have any history of serious adverse reactions to vaccines or drugs, such as allergy, urticaria, skin eczema, dyspnea, angoneeurotic edema, etc., which are deemed unsuitable for inclusion by researchers;
4. Patients with acute diseases or acute episodes of chronic diseases within 3 days before vaccination;
5. Before enrollment, the interval between other inactivated vaccines was less than 7 days, and the interval between live attenuated vaccines was less than 14 days;
6. Fever or antipyretic analgesics and antiallergic drugs were used in the first 3 days before enrollment;
7. Long-term use of immunosuppressants or other immunomodulatory drugs within 3 months prior to enrollment (defined as continuous use for more than 14 days), such as glucocorticoid dose ≥0.5mg/kg/ day (inhalation and local glucocorticoid are not restricted);
8. Received blood or blood related products 6 months before enrollment;
9. have been diagnosed with congenital or acquired immunodeficiency;
10. done with may interfere with study or severe disease or congenital malformations (including but not limited to, the researchers determine unfavorable into groups: respiratory diseases such as asthma or chronic bronchitis attack, down syndrome, during the Mediterranean anemia, heart disease, kidney disease, autoimmune diseases, genetic allergic constitution, GBS, skin diseases, etc.);
11. have been diagnosed with a systemic disease that may interfere with the conduct or completion of the study, such as tuberculosis, viral hepatitis, and/or human immunodeficiency virus HIV infection, as determined by the investigator to be ineligible for inclusion;
12. History or family history of convulsions, epilepsy, encephalopathy and mental illness;
13. There are contraindications to intramuscular injection, such as having been diagnosed with thrombocytopenia, any coagulation disorder or receiving anticoagulant treatment;
14. absence of spleen, functional absence of spleen, and absence of spleen or splenectomy resulting from any circumstance;
15. Plan to move out of the local area before the end of the study or leave the area for an extended period during the scheduled study visit;
16. The investigator considers that the subject has any conditions that might interfere with the evaluation of the study purpose.

The second dose delayed the standard of inoculation If any of the following occurs, the researchers will delay vaccination until the situation abates.

* Fever (axillary temperature ≥37.5℃ at visit);
* Acute illness or acute episode of chronic disease (within 3 days prior to vaccination);
* Insufficient interval between other vaccines (less than 7 days between inactivated vaccines and less than 14 days between live attenuated vaccines);
* Any other reasons that the investigator assessed to be necessary to delay trial vaccination.

Exclusion criteria for the second dose The investigator will discontinue the subject's trial vaccine if any of the following occurs.

* New discoveries or occurrences that meet the criteria for the first exclusion prior to vaccination (other than postponement of the criteria);
* Adverse reactions (including but not limited to) after vaccination (experimental vaccine);

appears within 48 hours after inoculation:

- High fever (axillary temperature ≥39.5°C), with or without convulsion;

appears after experimental vaccine is administered:

* encephalopathy;
* Seizures.

  * Other serious adverse events: decide whether to discontinue trial vaccine based on their treatment needs;
  * Any other reasons the investigator assessed to be necessary to discontinue trial vaccination.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Seroconversion Rate (SCR) | 28 days after the first dose of trial vaccine，30 days after the second dose of trial vaccine.
  Seroconversion Rate (SCR) of HI antibodies of 4 vaccine strain types in all subjects
Seroprotection Rate (SPR) | 28 days after the first dose of trial vaccine, 30 days after the second dose of trial vaccine.
  Seroprotection Rate (SPR) of HI antibodies of 4 vaccine types in all subjects
Geometric Mean Titer | 28 days after the first dose of trial vaccine，30 days after the second dose of trial vaccine.
  Geometric Mean Titer of HI antibodies of 4 vaccine types in all subjects
Incidence of adverse reactions | Incidence of adverse reactions within 0-28 (after the first dose) /0-30 (after the second dose) days after inoculation
  Incidence of adverse reactions within 0-28 (after the first dose) /0-30 (after the second dose) days after inoculation
Incidence of all adverse events | • Incidence of all adverse events 30 minutes after each dose;Incidence of all adverse events 7 days after each dose;
  • Incidence of all adverse events 30 minutes after each dose;Incidence of all adverse events 7 days after each dose;
Incidence of all serious adverse events | Incidence of all serious adverse events from the first dose to 6 months after full vaccination;
  Incidence of all serious adverse events from the first dose to 6 months after full vaccination;
Incidence of AE/SAE leading to withdrawal. | Incidence of AE/SAE leading to withdrawal within seven month during the study period
  Incidence of AE/SAE leading to withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Jikai Zhang, Principal Investigator — Guangdong province institute of biologicals and materia medica
Locations (1):
- Yangchun Center for Disease Control and Prevention, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
only for the objective of this study.